CLINICAL TRIAL: NCT06501274
Title: A Pragmatic Interventional Study to Assess the Clinical Value of Capsule Sponge in the Assessment of Response to Treatment of Non-stenotic Eosinophilic Oesophagitis in a Single District General Hospital
Brief Title: Capsule Sponge Study in Eosinophilic Oesophagitis
Acronym: Cosie
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD2022-43 314770
Record Dates: First submitted 2023-08-29; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Eosinophilic Esophagitis
Keywords: capsule sponge
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- all eligible patients with non stenotic eosinophilic oesophagitis (Other): single arm observational study
  Interventions: Device: capsule sponge

INTERVENTIONS:
Device: capsule sponge — capsule sponge sampling device of the oesophagus

SUMMARY:
Open pragmatic, descriptive single site study in adult patients with non-stenotic eosinophilic oesophagitis.

To assess the clinical value of Capsule sponge in the assessment of treatment response in patients with known non-stenosing eosinophilic oesophagitis, as an alternative to gastroscopy in a real world setting.

To assess patient preference for Capsule sponge or gastroscopy. All patients with non-stenosing eosinophilic oesophagitis who are reviewed in clinic that have not had reassessment of their oesophagus post treatment initiation or change in treatment will be offered Capsule sponge as an alternative to gastroscopy.

A standardised clinical symptom questionnaire will be self-administered for 2w prior to clinic visits and Capsule sponge.

Telephone triage for safety check and exclusion criteria by Capsule sponge nurse.

A patient symptom questionnaire at the time of procedure by research nurse. A patient satisfaction survey will be delivered after the Capsule sponge procedure by Capsule sponge nurse.

Cytological assessment of the Capsule sponge and eosinophil count and other markers of inflammation will be reported by Cyted.

Clinic follow up will occur at approximately 6-8 weeks post Capsule sponge. Descriptive Changes in management as a result of the Capsule sponge findings and /or symptoms will be recorded by clinician.

DETAILED DESCRIPTION:
Eosinophilic oesophagitis is a condition characterised by symptoms of dysphagia (swallowing difficulties) and/or food impaction in adults, with oesophageal biopsies (histology) showing a peak eosinophil count of >15 eosinophils/high power field (or >15 eosinophils/0.3mm2 or >60 eosinophils / mm2), and the absence of other causes of oesophageal.

Evidence suggests that if inadequately treated there is increased risk of oesophageal fibrosis and stricture formation that can lead to progressive dysphagia, food bolus obstruction (food blockages) and increased morbidity. The degree of eosinophil infiltration in the mucosa is thought to reflect the disease activity better than patient symptoms.

Current guidelines from Europe and newly published national guidelines from the British Society of Gastroenterology from the UK recommend reassessment of oesophageal eosinophilia after treatment to ensure remission This has traditionally involved repeating gastroscopies after each treatment (diet -after each food group, proton pump inhibitor (PPI), topical steroids) which is unpleasant for patients, expensive and labour intensive as well as producing a large carbon footprint.

Since the start of the COVID-19 pandemic in January 2020 there has been restricted or delayed access to gastroscopy nationally and consequently many patients with EOE have had their repeat gastroscopies cancelled or postponed, increasing the risk of complications from undertreated disease.

Capsule sponge (Cytosponge and Endosign being the current commercially produced example in the UK) is an oesophageal cell sampling device that is a 'pill on a string'. The patient swallows the pill with water and the sponge expands in the stomach. The nurse withdraws the string after 7 minutes and the sponge collects oesophageal cells on withdrawal. The sponge is sent for cytological analysis that identifies cells that can be stained for various biomarkers of Barrett's oesophagus (TFF3) and markers of dysplasia (p53 and atypia) as well as the opportunity to look at inflammation and in particular in this setting to assess the number of eosinophils and other histological and inflammatory markers supporting a diagnosis of EOE.

The use of Capsule sponge in the diagnosis and monitoring of EOE has been described as an alternative to gastroscopy and a quantitative eosinophil count is possible on cytology to allow sequential assessment. The eosinophil count on cytology samples from Capsule sponge are similar to biopsies taken from the same patient at the same time, when assessed per high power field (area of 0.3mm2) in a single study.

Over 10,000 Capsule sponge procedures have now been performed in the UK. The Capsule sponge service at East and North Herts trust has now performed over 1000 procedures making the trust the largest UK single site experience.

The trial population will involve adult patients over 18 years who are known to have a histological diagnosis of EOE and are under follow up at East and North Herts NHS trust.

Preclinical/Clinical Data The use of Capsule sponge in the monitoring of EOE has been described in a single prospective cross sectional 2-centre study in USA .

There have been no studies to date assessing the clinical value of Capsule sponge in monitoring disease activity or response to treatment in adults in a real-world setting.

Rationale

* Does the use of Capsule sponge instead of endoscopy and biopsies in monitoring known non-stenotic EOE provide sufficient information to affect management decisions in a real-world setting?
* Current practice to monitor EOE disease activity with endoscopy and biopsies has been severely affected by the COVID19 pandemic resulting in delays to treatment and the risk of progressive stenotic disease and morbidity.
* Gastroscopy is invasive, expensive, unpleasant and aerosol generating whilst Capsule sponge is cheaper, much less invasive does not require sedation and is preferred by patients and carries a lower carbon footprint.

STUDY OBJECTIVES AND DESIGN Objectives Primary objectives: Does Capsule sponge instead of endoscopy and biopsies in monitoring known non stenotic EOE provide sufficient information to affect management decisions in a real-world setting? Do patients show a preference for Capsule sponge over endoscopy and biopsies?

Secondary objectives:

* Subgroup analysis by current treatment
* Do Symptom scores reflect eosinophil count and other markers of inflammation on cytology and histology?
* Complications
* Failure to swallow rate
* Inadequate cytology rate
* Gastroscopy rate by 1year if not done simultaneously
* Potential Cost savings compared with gastroscopy

Endpoints/outcomes

Primary Endpoints/outcomes:

Descriptive analysis of management decision made as a result of the Capsule sponge findings Patient preference for Capsule sponge or gastroscopy

Secondary Endpoints/outcomes:

* Subgroup analysis by current treatment (diet/PPI/topical steroid/combination/no treatment)
* Correlation between Symptom scores and eosinophil count and other markers of inflammation on cytology and histology
* Additional cytological findings of EOE activity and inflammation
* Other cytological findings: Barrett's oesophagus/dysplasia/other diagnoses
* Number of Complications
* Failure to swallow rate
* Inadequate cytology rate
* Gastroscopy rate if not done simultaneously
* Cost savings
* Patient satisfaction and pain scores

Study Design

* Purpose of research To identify a suitable alternative to endoscopic biopsies for monitoring patients with non-stenotic EOE.
* Real-world prospective pragmatic interventional study in a single district general hospital secondary care setting with quantitative and qualitative outcome measures. Design chosen as pragmatic and comparative control study with endoscopy would be impractical due to COVID backlog, cost and such a study has already been performed
* Data collection methods:
* An excel database of patients with EOE will be established and used as a screening log.

With demographic data, date of diagnosis, date of previous endoscopies, endoscopic findings (EREFS criteria if documented) eosinophil count on previous histology and any other histological supportive features, current and previous treatments documented. Reasons for ineligibility will also be documented.

The study will be discussed with eligible patients at their normal clinic appointment and for eligible patients who agree to enrol in the study:

The following will be sent to patient by email/post as preferred and the Capsule sponge service contact email and phone details:

* Eligible patients will be sent copies of the trust standard Capsule sponge procedure information leaflet.
* Copies of patient Information leaflet regarding the COSiE trial
* Study specific Consent form
* 2 week symptoms diary Dysphagia Symptom Questionnaire (DSQ)

The following will be administered with the patient on the day of the Capsule sponge procedure:

* Capsule sponge eligibility and safety questionnaire
* Documentation of Current treatment and duration and compliance
* Patient satisfaction survey after procedure

Patient participation opinion group has been completed

Number of subjects A total of 100 -140 evaluable patients will be enrolled in the study. This is thought to be an achievable sufficiently large sample target given the prevalence of EOE in the catchment population. The PI runs a dedicated EOE teleclinic every month that sees approximately 12 patients. It is estimated that 2/3 of these would be eligible for Capsule sponge. In addition, other patients with EOE are also followed up in 5 other consultant gastroenterology clinics that would be eligible for the study.

Study Duration The length of time the study is expected to run over 2 years in order to recruit sufficiently large sample.

ELIGIBILITY:
Inclusion Criteria:

• patients diagnosed with non -stenotic eosinophilic oesophagitis who have a change in treatment

Exclusion Criteria:

* Strictures or rings at most recent endoscopy that prevent passage of adult gastroscope
* Previous oesophageal dilatation
* Previous oesophageal perforation or surgical resection
* Oesophago-gastric malignancy
* Oesophageal varices
* Bolus obstruction since last endoscopy requiring hospital visit
* Previous fundoplication or complicated hiatus hernia
* Patient on Warfarin with INR>=3
* Suspected new diagnosis of EOE without prior endoscopic confirmation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
• Descriptive Changes in clinical management of EOE following Capsule sponge assessment | through study completion, an average of 1 year
  has the results of the capsule sponge resulted in a decision to change treatment drug, or drug dose?-yes/ no response
• symptom score | through study completion, an average of 1 year
  Dysphagia symptom score (DSQ) scored as continuous variable in 2 weeks prior to capsule sponge
• Eosinophil count on cytology | through study completion, an average of 1 year
  no of eosinophils per high powered field on cytology
• Patient pain evaluation | through study completion, an average of 1 year
  wong -baker faces visual scale from 0 to 10 with 0 being no pain and 10 being maximum pain
patient preference for endoscopy or capsule sponge | through study completion, an average of 1 year
  tick box

SECONDARY OUTCOMES:
• Failure to swallow rate | through study completion, an average of 1 year
  proportion of patients unable to swallow device after 2 attempts
• Inadequate sample rate | through study completion, an average of 1 year
  proportion of samples with inadequate squamous cells for analysis
• Complications | through study completion, an average of 1 year
  recognised immediate complications
• Repeat gastroscopy rate | through study completion, an average of 1 year
  numbers of patients requiring gastroscopy within 1year of sponge
Cost evaluation | at end of study at 2 years
  comparison of sponge v gastroscopy real world costs of service in GB Pounds

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Morris, MD FRCP, Principal Investigator — East and North Herts NHS Trust
Locations (1):
- East and North Herts NHS Trust, Stevenage, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
there is no current plan to make de-identified individual participant data (IPD) collected in this study available to other researchers (e.g., outside the primary research group). Individual requests for data sharing can be considered on request via email

REFERENCES:
- [Background] Dhar A, Haboubi HN, Attwood SE, Auth MKH, Dunn JM, Sweis R, Morris D, Epstein J, Novelli MR, Hunter H, Cordell A, Hall S, Hayat JO, Kapur K, Moore AR, Read C, Sami SS, Turner PJ, Trudgill NJ. British Society of Gastroenterology (BSG) and British Society of Paediatric Gastroenterology, Hepatology and Nutrition (BSPGHAN) joint consensus guidelines on the diagnosis and management of eosinophilic oesophagitis in children and adults. Gut. 2022 Aug;71(8):1459-1487. doi: 10.1136/gutjnl-2022-327326. Epub 2022 May 23. PMID 35606089
- [Background] di Pietro M, Modolell I, O'Donovan M, Price C, Pilonis ND, Debiram-Beecham I, Fitzgerald RC. Use of Cytosponge as a triaging tool to upper gastrointestinal endoscopy during the COVID-19 pandemic. Lancet Gastroenterol Hepatol. 2020 Sep;5(9):805-806. doi: 10.1016/S2468-1253(20)30242-9. Epub 2020 Jul 30. No abstract available. PMID 32738939
- [Background] Paterson AL, Lao-Sirieix P, O'Donovan M, Debiram-Beecham I, di Pietro M, Miremadi A, Attwood SE, Walter FM, Sasieni PD, Fitzgerald RC; BEST and BEST2 study groups. Range of pathologies diagnosed using a minimally invasive capsule sponge to evaluate patients with reflux symptoms. Histopathology. 2017 Jan;70(2):203-210. doi: 10.1111/his.13039. Epub 2016 Oct 12. PMID 27417524
- [Background] Katzka DA, Smyrk TC, Alexander JA, Geno DM, Beitia RA, Chang AO, Shaheen NJ, Fitzgerald RC, Dellon ES. Accuracy and Safety of the Cytosponge for Assessing Histologic Activity in Eosinophilic Esophagitis: A Two-Center Study. Am J Gastroenterol. 2017 Oct;112(10):1538-1544. doi: 10.1038/ajg.2017.244. Epub 2017 Aug 15. PMID 28809387
- [Background] Januszewicz W, Tan WK, Lehovsky K, Debiram-Beecham I, Nuckcheddy T, Moist S, Kadri S, di Pietro M, Boussioutas A, Shaheen NJ, Katzka DA, Dellon ES, Fitzgerald RC; BEST1 and BEST2 study investigators. Safety and Acceptability of Esophageal Cytosponge Cell Collection Device in a Pooled Analysis of Data From Individual Patients. Clin Gastroenterol Hepatol. 2019 Mar;17(4):647-656.e1. doi: 10.1016/j.cgh.2018.07.043. Epub 2018 Aug 9. PMID 30099104
- [Background] Swart N, Maroni R, Muldrew B, Sasieni P, Fitzgerald RC, Morris S; BEST3 Consortium. Economic evaluation of Cytosponge(R)-trefoil factor 3 for Barrett esophagus: A cost-utility analysis of randomised controlled trial data. EClinicalMedicine. 2021 Jun 18;37:100969. doi: 10.1016/j.eclinm.2021.100969. eCollection 2021 Jul. PMID 34195582
- [Background] Hudgens S, Evans C, Phillips E, Hill M. Psychometric validation of the Dysphagia Symptom Questionnaire in patients with eosinophilic esophagitis treated with budesonide oral suspension. J Patient Rep Outcomes. 2017;1(1):3. doi: 10.1186/s41687-017-0006-5. Epub 2017 Sep 12. PMID 29757322
- [Background] Dellon ES, Irani AM, Hill MR, Hirano I. Development and field testing of a novel patient-reported outcome measure of dysphagia in patients with eosinophilic esophagitis. Aliment Pharmacol Ther. 2013 Sep;38(6):634-42. doi: 10.1111/apt.12413. Epub 2013 Jul 9. PMID 23837796